CLINICAL TRIAL: NCT04301206
Title: Videos and Simple Text to Empower Parents to Handle Their Sick Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emergency Medical Services, Capital Region, Denmark (Other Government)
Collaborators: Copenhagen University Hospital, Hvidovre (Other); Copenhagen University Hospital at Herlev (Other); Rigshospitalet, Denmark (Other); University Hospital Bispebjerg and Frederiksberg (Other); Hospital of Bornholm, Denmark (Unknown); University of Copenhagen (Other); Copenhagen University Hospital Nordsjælland (Unknown); TrygFonden, Denmark (Industry); Region Headquarters, Copenhagen (Regionsgården, Region Hovedstaden) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: BB
Record Dates: First submitted 2020-02-26; First posted 2020-03-10 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Pediatrics; Efficacy, Self; Triage
Keywords: education in medical conditions

STUDY DESIGN:
Intervention Model Description: The parents of children aged 6 months to 11.9 years who calls 1813 about a medical condition will be offered to participate in the study. They will hear a recorded instruction, explaining the study. If they accept to participate they will be allocated to the intervention group and the control group 1:1.
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Receiving video material (Experimental): The parents who accepts to participate and receives videos and action cards by sms
  Interventions: Behavioral: Intervention Group
- Control group (No Intervention): The parents who accepts to participate, but proceed to 1813 and do not receive videos and action cards

INTERVENTIONS:
Behavioral: Intervention Group — Empowerment of parents. When calling the medical helpline 1813 the parents will be offered to access the new material about sick children, compared to not getting this possibility.
  Arms: Intervention: Receiving video material

SUMMARY:
Background:

The Medical Helpline 1813 (Capital Region, Denmark) handles acute, non-life-threatening medical emergencies. Approx. 200,000 calls/year concern children (ref: Rasmussen et al), and about 30% are referred to a pediatric urgent care center. However, many of these children presents very mild symptoms, which require neither treatment nor paraclinical tests, merely parental guidance.

We want to empower the parents when handling their sick children by videos and simple text accessible from their smartphone. We want the parents to handle mild symptoms at home and to know when they must contact the medical helpline 1813 or a general practitioner.

We have produced 8 short videos and simple texts about the most common symptoms in sick children. The material covers about 70% of the symptoms in acute sick children. The material is developed in collaboration between pediatricians and professional movie producers and is approved by the Danish Society of Pediatrics and other relevant medical societies.

Purpose:

It will be studied if the new material about symptoms in sick children result in 5% higher parental self-efficacy among the parents who were allowed to watch the material.

Moreover, it will be studied if the new material resulted in less children examined by a doctor, and satisfied parents.

Method:

Parents who call the medical helpline about a medically ill child aged 6 months to 12 years will be offered to try the new material. If they accept, every second parent will be allowed given access to the new material, and every other parent will receive the usual triage by telephone. The results of these otherwise similar groups will be compared. Parents answer surveys about their experiences.

Yield:

Videos and simple text may empower parents to handle their sick children. The study may result in fewer children referred to hospitals, more appropriate use of resources and better experiences for the families.

DETAILED DESCRIPTION:
Background:

Each year there are approximately 200.000 calls regarding sick children younger than 12 years (injuries excluded) to the medical helpline 1813 in the Capital Region of Denmark (ref: Rasmussen et al). These children are not so ill that the parents call the emergency helpline 112, but the parents need to contact the health care system outside their general practitioners' opening hours. After contact with the parents, the medical helpline health professionals (primarily physicians or nurses) may either: 1) refer the child to a pediatric department, 2) refer child to assessment in a pediatric urgent care center, 3) guide the parents on how to perform self-care at home or 4) advice the child to the general practitioners next work day. About 40 % of the calls to 1813 regarding children are referred to a hospital. We estimate that 40 % of those presents mild symptoms, which often does not require treatment or paraclinical tests and many could have benefitted from being observed at home.

Purpose:

Reviews conducted in child health related areas, have indicated that quality of health information varies significantly and Internet searches may reveal information that is not evidence-based, or may even be inconsistent with international treatment recommendations (ref: Pehora et al, Fahy et al). Often health information will also focus on diagnosis, not symptoms, which makes it difficult for parents to navigate the health directions. The study objective is to investigate if it is possible by using videos and simple action cards about common symptoms in children - to empower parents and citizens to take better care of sick children with milder symptoms at home including to know when they must call for medical help. This project therefore aims to, by increasing parental knowledge, decrease the number of children admitted to the hospital with mild symptoms, and to decrease the number of children with late arrival to the hospital with symptoms on critical illness.

Method:

Eight videos have been produced, each lasting about 2-3 minutes, about the following common symptoms: 1) vomiting or diarrhea, 2) difficulties in breathing, 3) fever, 4) abdominal pain, 5) sore throat, 6) a red eye, 7) pain in the ears, and 8) exanthemas. The videos will be accompanied by text, action cards, and be accessible on a smartphone. The information is in Danish. The material has been developed in collaboration between pediatricians (medical content) and professional film/app-makers (creative content) and has been approved by the Danish Society of Pediatrics and other relevant scientific societies. We want to study the clinical value of this material before we launch the campaign to the public.

Parents with children aged between 6 months - 11.9 years will, when contacting the medical helpline 1813, be offered to receive a new information material. If they accept, they will be randomized to the intervention group (randomized to the new material composed of 8 videos and corresponding smart cards) or to the control group (randomized to current standard care). The participants will the following day receive a text message with six questions on self-efficacy and satisfaction. If the caretaker does not fill out the electronical questionnaire, they will receive a reminder the next day. All case reports of the included children will be reviewed and if admitted to a hospital in the Capital Region of Denmark within 72 hours of the call, the diagnosis, duration and treatment will be registered. For the intervention group, the use of the material will be logged.

Statistics:

The primary analysis will use Chi-square and a two-sided level of significance of p < 0.05 for the primary outcome and a p<0.025 for the two secondary outcomes. All other outcomes are exploratory and the statistical methods will be adapted as appropriate. The results from these exploratory analyses will not but used to claim clinical efficacy but used to design new studies. This is an important aspect since new studies can be rapidly designed and performed once the project set-up is in place.

Sample size:

We want to be able to detect if the intervention with videos and action cards increases the proportions of parents who expressed high self-efficacy by 5%. We do not know this actual proportion. If it is actually 50%, we want to detect an increase to 55%. We want a p-value of 0.05 and a probability (power) of 80%. It will require data from about 3300 text-messages in total, randomized in two equal groups (http://www.openepi.com/SampleSize/SSCohort.htm). We suggest we have data to answer our research question within 3 months, and the study will be stopped after 6 months.

After the first 400 SMS-answers, we will perform an interim analysis to study the frequency of acceptance, and the frequency of high self-efficacy, as well as how the videos have worked technically. Moreover, we will study if the number of SMS-answers from the two groups of families, those randomized to intervention and those randomized to control, are about the same size.

After the first 1000 SMS-answers, we will also make an interim analysis to study the effect of the videos and the action cards. This will also include an examination of a significant difference is exhibited between the number of children staying at home the day the parents call 1813 after having the possibility to watch the videos and read the action cards.

Ethics and transparency:

The parents are informed about the study by an automatic voice message when contacting the medical helpline 1813. Their acceptance to the study is their informed consent. The project will be described in short at the webpage of the Copenhagen Emergency Service, where it will be possible to access additional information via a link to the study at Clinical Trials. The telephone call will be recorded in the Emergency Medical Services system, based on the actual regular routine. The protocol has been submitted to the Ethics Committee of the Capital Region of Denmark, who considered it outside their mandate.

In the project the data will be completely anonymized and it is in no way possible to link data with actual people. The study will be registered at https://clinicaltrials.gov/ before enrolment of the first patient.

In cases of serious adverse events the study group will consider stopping the study. This will also be the case if the satisfaction with the contact to the medical helpline 1813 drops to a very low level.

Perspectives and possible yield:

In case of positive effect, it must be decided if the videos and action cards will be an integrated option at the medical helpline 1813. Moreover, it may be considered if the material is released to all of Denmark. The material could be accessible at smartphones, iPads, laptops and easy to find on different major national websites.

ELIGIBILITY:
Inclusion Criteria:

* Parents calling 1813 with children aged 6 months to 11,9 years who accepts to receive the new information material.

Exclusion Criteria:

* Children with parents who do not speak Danish
* Children without a Danish civil registration number
* The parent does not call from a Danish number
* Parents calling 1813 with children with an injury
* Parents calling 1813 within 72 hours regarding same child
* Parents who are not calling from a smart-phone

Ages: 6 Months to 143 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1558 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Changed in parental self-efficacy: Difference in the number of parents in the two arms suggesting that the new material about sick children resulted in an changed parental self-efficacy among the parents who were allowed to watch the material | the parents are sent a link to an online questionnaire at 12pm the day after the medical helpline contact
  Difference in the number of parents in the two arms suggesting that the new material about sick children resulted in an changed parental self-efficacy among the parents who were allowed to watch the material. High parental self-efficacy defined as parents who answered "very much" or "to a great extent" to at least two of the following questions:
  "To which degree were you able to take care of your child, after contacting 1813?" "Do you know what to do at home, if your child presents the same symptoms another time?" "Do you know, the critical point at which you should contact your GP or 1813, if your child develops the same symptoms another time?"

SECONDARY OUTCOMES:
Use of professional consultations | Registered by questionnaire sent out at 12pm the day after the medical helpline contact
  Difference in the number of parents in the two arms who answered Yes to the question "Did a nurse/doctor examine your child during this period of sickness?"
Did the new material about sick children result in more satisfied parents? | Registered by questionnaire sent out at 12pm the day after the medical helpline contact
  Difference in the number of parents in the two arms who expressed a "very high degree" or "high degree" of satisfaction
Course of action at the medical helpline | disposition is registered by the call operator immediately after the call
  Difference between the two arms in the percentage of children that are given health-information, performing video transmission for telephone triage, using the "call-back"- option , administrating any sort of treatment during the medical helpline-call, admission to hospital, ambulance, doctors ambulance
Hospital visits | the hospital chart of all children are read within 3-8 days after the call
  difference between the two arms in the percentage of how many children that are seen at a hospital within 8 hours hours, 12 hours, 24 hours, 48 hours, 48-72 hours after the call to medical helpline, and does that match the disposition registered by the medical professional at the medical helpline? Which diagnosis was given at the hospital? If admitted to the hospital, are there then any difference between the two arms in the percentage of how many children received treatment and paraclinical test? If admitted to the hospital, are there then any difference between the two arms in the percentage of the duration and type of admission?
Non-participating parents | these parameters will be studied at the completion of enrollment of patients
  Description of differences in the ages, diagnoses, dispositions between the children whose parents wanted to participate in video triage and those who did not.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Cortes, MD, DrMedSci, Study Chair — Department of Pediatrics, Copenhagen University Hospital Hvidovre
Locations (1):
- Emergency Medical Services, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rasmussen, MV. Sektionen for data, controlling og IT, Akutberedskabet, Region Hovedstaden. January 2018 (data extract from the patient database at Emergency Services, Copenhagen)
- [Background] Pehora C, Gajaria N, Stoute M, Fracassa S, Serebale-O'Sullivan R, Matava CT. Are Parents Getting it Right? A Survey of Parents' Internet Use for Children's Health Care Information. Interact J Med Res. 2015 Jun 22;4(2):e12. doi: 10.2196/ijmr.3790. PMID 26099207
- [Background] Fahy E, Hardikar R, Fox A, Mackay S. Quality of patient health information on the Internet: reviewing a complex and evolving landscape. Australas Med J. 2014 Jan 31;7(1):24-8. doi: 10.4066/AMJ.2014.1900. eCollection 2014. PMID 24567763
- [Derived] Borch-Johnsen L, Gren C, Lund S, Folke F, Schroder M, Frederiksen MS, Lippert F, Ersboll AK, Greisen G, Cortes D. Video Tutorials to Empower Caregivers of Ill Children and Reduce Health Care Utilization: A Randomized Clinical Trial. JAMA Netw Open. 2023 Oct 2;6(10):e2336836. doi: 10.1001/jamanetworkopen.2023.36836. PMID 37824145

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT04301206/Prot_SAP_000.pdf